CLINICAL TRIAL: NCT03123835
Title: Outcome Analysis of Endoluminal Therapies for Gastrointestinal Conditions Compared to Current Treatment Paradigms
Brief Title: Outcome Analysis of POEM and Endoluminal Therapies
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 676956
Record Dates: First submitted 2016-04-05; First posted 2017-04-21 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Achalasia; Gastric Fistula; Weight Gain After Primary Weight Loss Surgery; Marginal Ulcer; Stenoses; Gastric Nec
Keywords: Achalasia; Fistula; Obesity; POEM; GERD; endoscopic; treatments; post bariatric surger weight gain; endoluminal; Bariatric Surgery; Barretts
MeSH Terms: conditions — Esophageal Achalasia; Gastric Fistula; Peptic Ulcer; Constriction, Pathologic; Fistula; Obesity; Gastroesophageal Reflux | interventions — nephronectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other): Patients meeting inclusion criteria for possible surgical therapies for their current condition (IE Achelasia, Enlarged Gastric Pouch and/or Gastrogastric Fistula after primary weight loss surgery, etc) will be educated on the different therapy options including traditional laparoscopic surgery and/or Endoscopic Interventions including POEM (Percutaneous Oral Endoscopic Myomectomy for the treatment of Achelasia) or Endoscoscopic Pouch/GastroJejunostomy repair or closure of the Gastrogastric Fistula as examples.
  Interventions: Procedure: Endoscopic Intervention

INTERVENTIONS:
Procedure: Endoscopic Intervention — After reviewing all therapeutic options the patient will be offered the best therapeutic option to treat their condition. Surgical interventions include open laparotomy, diagnostic/therapeutic laparoscopy or endoluminal therapies. After the patient is consented for the related surgical intervention the patient will be given the option to participate in the clinical study to measure outcomes after surgery.
  Other Names: Endoluminal Therapies, POEM, Endoscopic Revision

SUMMARY:
Evaluation of current and newly developed endoluminal therapies in the management of Upper and Lower GI conditions.

DETAILED DESCRIPTION:
Over the last few years there have been numerous advances in the use of endoscopic equipment and related treatments in the identification and intervention of gastrointestinal diseases. Many of these treatments using flexible endoscopes have either complimented or replaced surgical approaches to these same benign and malignant disease processes with the potential of being the standard of care for many of these clinical conditions. The initial primary focus of this study will be the use of endoscopic myotomy for achalasia, endoscopic treatment of post bariatric weight gain, endoscopic gastro-gastric fistula treatments, and other endoluminal therapies for gastrointestinal and post-operative conditions. These treatments have been validated by prior surgery studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients 18-80 years of age
* Meet the criteria for surgery of benign and/or malignant gastrointestinal pathology(s)
* Gastrointestinal Reflux Disease
* Achalasia
* Barrett's Esophagus
* Post Bariatric Surgery conditions
* Other gastrointestinal and postsurgical disorders.

Exclusion Criteria:

* Adults unable to consent
* Individuals that do not meet inclusion criteria or qualify for endoluminal treatment paradigms and internees.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-03; Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Decrease in GERDDQ | 3-6 months
  Assessment will be made via post surgery questionnaire (decreasing in scoring will be 0-5)

SECONDARY OUTCOMES:
Decrease in Eckardt scoring | 30 days
  Decrease in overall GERD symptoms using Eckardt Scoring methodology (5-0)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R Ali, MD, Principal Investigator — U.C. Davis Medical Center
Locations (1):
- Univesity of California Davis Health System, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
de-identified data will be maintained until study closure. Statistical summary of data will be published with any journal articles submitted for review/approval.